CLINICAL TRIAL: NCT05340647
Title: NorMIGS - a Prospective Study of Micro-invasive Glaucoma Surgery
Brief Title: NorMIGS - a Study of Micro-invasive Glaucoma Surgery
Acronym: NorMIGS
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Olav Kristianslund, Principal investigator, Head of section / Senior consultant MD PhD, Oslo University Hospital
Other Study IDs: 415116
Record Dates: First submitted 2022-04-09; First posted 2022-04-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 Preserflo microshunt
  Interventions: Procedure: Preserflo microshunt
- Group 2 Trabeculectomy
  Interventions: Procedure: Trabeculectomy
- Group 3 Other MIGS: Other micro-invasive glaucoma surgery (MIGS) than Preserflo microshunt (e.g., Xen gel stent, iStent inject)
  Interventions: Procedure: Other MIGS

INTERVENTIONS:
Procedure: Preserflo microshunt — Implantation of Preserflo microshunt (Santen) to lower intraocular pressure
  Groups: Group 1 Preserflo microshunt
Procedure: Trabeculectomy — Trabeculectomy surgery to lower intraocular pressure
  Groups: Group 2 Trabeculectomy
Procedure: Other MIGS — Other MIGS than Preserflo microshunt (e.g., XEN gel stent, iStent inject) to lower intraocular pressure
  Groups: Group 3 Other MIGS

SUMMARY:
NorMIGS is a non-randomized clinical study of intraocular pressure lowering effect and complications after Preserflo microshunt implantation versus other types of glaucoma surgery. The study is conducted in the Department of Ophthalmology, Oslo University Hospital, Norway.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older at the time of signing the informed consent form. There is no upper age limit.
* Scheduled for implantation of Preserflo microshunt, trabeculectomy or other types of MIGS
* Ability to cooperate fairly well during the examinations
* Willing to participate in the study and capable of providing informed consent

Exclusion Criteria:

- High intraocular pressure due to increased episcleral venous pressure, hemorrhagic glaucoma, traumatic glaucoma or uveitis glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients referred to the Department of Ophthalmology, Oslo University Hospital, for glaucoma surgery. The operation type will be decided by clinicians regardless of study participation, and they will be assigned to study groups based on this clinical decisions (non-interventional). In addition, the type of glaucoma will be determined, which is relevant for sub group analyses (pseudoexfoliation groucoma (PEXG), primary open-angle glaucoma (POAG) and other types).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 8 weeks after surgery
  Measured by tonometry

SECONDARY OUTCOMES:
Intraocular pressure | 6 months after surgery
  Measured by tonometry
Intraocular pressure | 2 years after surgery
  Measured by tonometry
Intraocular pressure | 5 years after surgery
  Measured by tonometry
Visual outcome | 8 weeks after surgery
  Measure uncorrected and corrected distance visual acuity using visual acuity chart
Visual outcome | 6 months after surgery
  Measure uncorrected and corrected distance visual acuity using visual acuity chart
Visual outcome | 2 years after surgery
  Measure uncorrected and corrected distance visual acuity using visual acuity chart
Visual outcome | 5 years after surgery
  Measure uncorrected and corrected distance visual acuity using visual acuity chart
Intraocular inflammation | 4 weeks after surgery
  Measured by laser flare meter
Intraocular inflammation | 6 months after surgery
  Measured by laser flare meter
Central macular thickness (CMT) | 4 weeks after surgery
  Measure CMT (in um) on optical coherence tomography (OCT)
Central macular thickness (CMT) | 6 months after surgery
  Measure CMT (in um) on optical coherence tomography (OCT)
Corneal endothelial cell density | 6 months after surgery
  Measured by confocal or spectral microscopy
Corneal endothelial cell density | 2 years after surgery
  Measured by confocal or spectral microscopy
Corneal endothelial cell density | 5 years after surgery
  Measured by confocal or spectral microscopy
Patient reported outcome measure (PROMs) | 6 months after surgery
  EuroQol-5 D (EQ-5D) questionnaire
Patient reported outcome measure (PROMs) | 2 years after surgery
  EuroQol-5 D (EQ-5D) questionnaire
Patient reported outcome measure (PROMs) | 6 months after surgery
  National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ 25)
Patient reported outcome measure (PROMs) | 2 years after surgery
  National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ 25)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Kristianslund, MD PhD, Principal Investigator — Department of Ophthalmology, Oslo University Hospital
Locations (1):
- Department of Ophthalmology, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided